CLINICAL TRIAL: NCT05831462
Title: Standard Versus Low Dose Maintenance Ticagrelor After Primary Percutaneous Intervention for STEMI in Diabetic Patients: a Randomized Controlled Trial
Brief Title: De-escalation of Ticagrelor in Post PPCI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Taha Galal, Cardiology specialist at assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ticagrelor in post PPCI
Record Dates: First submitted 2023-02-18; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Ticagrelor
Keywords: post- PPCI
MeSH Terms: interventions — Ticagrelor

STUDY DESIGN:
Intervention Model Description: cvbnm-89
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard dose ticagrelor with aspirin in patients post PPCI for 1 year. (Active Comparator): Drug: Ticagrelor 90 mg until 1 year after PPCI (other name: Brillique). Drug: Aspirin 75 mg until 1 year after PPCI.
  Interventions: Drug: Ticagrelor 60mg
- Low-dose Ticagrelor with aspirin in patients post PPCI (Experimental): Patients will recieve the following antiplatlet therapy:
  1. Ticagrelor 2x90 mg + aspirin 1x 75 during the first three months post PPCI.
  2. Ticagrelor 2x60 mg + aspirin 1x 75 after the first three months post PPCI until one year post PPCI.
  Interventions: Drug: Ticagrelor 60mg

INTERVENTIONS:
Drug: Ticagrelor 60mg — Standard vs Low dose ticagrelor in post PPCI patients
  Other Names: Brillique

SUMMARY:
Primary objective: to evaluate the efficacy and safety of De-escalation to lower dose Ticagrelor (60 mg BID) plus Aspirin (75 mg OD) versus continuation of standard dose Ticagrelor (90 mg BID) plus Aspirin (75 mg OD), 1 month after primary PCI for STEMI, in diabetic patients.

Secondary objectives:

To compare tolerability and discontinuation of Ticagrelor in both doses. To compare the 1ry safety & efficacy endpoints in subgroups with different thrombotic/ischemic risk

DETAILED DESCRIPTION:
[15:42, 18/02/2023] M Taha: Ticagrelor at a maintenance dose of 90 mg twice a day (bid) was shown to provide greater and more consistent platelet P2Y12 inhibition than clopidogrel in patients with stable coronary artery disease (PA Gurbal, KP Bliden et al 2009) and acute coronary syndromes (ACS) (RF Storey, S Husted et al 2007).

The PLATO (Platelet Inhibition and Patient Outcomes) trial demonstrated the superior efficacy of ticagrelor, given at a maintenance dose of 90 mg bid, compared with clopidogrel for up to 1 year in patients with ACS (L Wallentin, RC Becker et al 2009) [15:42, 18/02/2023] M Taha: Consequently, this regimen of ticagrelor is recommended in international guidelines as first-line therapy for up to 1 year following either non-ST-segment elevation ACS (P Damman, AW van't Hof et al 2017) or ST-segment elevation myocardial infarction managed with primary percutaneous coronary intervention (PT O'gara, FG Kushner et al 2013).

In the PEGASUS-TIMI 54 trial, ticagrelor maintenance doses of 60 mg b.i.d and 90 mg b.i.d were clinically equally effective in stable patients more than 1 year after acute myocardial infarction (AMI), with a better tolerability of treatment observed with the lower dose (Bonaca MP, Bhatt DL et al 2016).

[15:42, 18/02/2023] M Taha: n a pharmacokinetic & pharmacodynamic substudy of the PEGASUS-TIMI 54 trial, ticagrelor 60 mg bid achieved high levels of peak and trough platelet inhibition in nearly all patients, similar to that with 90 mg bid, helping to explain the efficacy of the lower ticagrelor dose in the trial.1 Most recently, in a pharmacodynamic randomized controlled study (ELECTRA), lowering ticagrelor maintenance dose to 60 mg b.i.d, on day 30 following acute MI, was shown to confer an adequate antiplatelet effect that is comparable to the standard maintenance dose of 90 mg b.i.d.2

ELIGIBILITY:
Inclusion Criteria:

Diabetes Mellitus. Acute STEMI. Able to swallow tablets.

Exclusion Criteria:

Patients presenting with stent thrombosis. Hypersensitivity to ticagrelor and/or aspirin. Active bleeding. ARC-high bleeding risk status1. 2nd or 3rd degree AV block. Previous stent thrombosis on treatment with ticagrelor. Pregnancy or lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
primary efficacy endpoint, primary safety endpoint | after 12 months
  including CV death, non-fatal MI, non-fatal stroke, coronary revascularization barc 2,3,5 bleeding

SECONDARY OUTCOMES:
secondry endpoints | after 12 months
  dyspnea leading to discontinuation of ticagrelor, barc 1 bleeding leading to discontinuation of the drug

REFERENCES:
- See also: Related Info — http://journals.sagepub.com/doi/pdf/10.1177/0003319716674855
- See also: Related Info — http://journals.viamedica.pl/cardiology_journal/article/view/84307